CLINICAL TRIAL: NCT04400721
Title: The Effects of Thoracic Nerve Blocks on Postoperative Pain, Respiratory Function and Recovery in Patients Undergoing Thoracoscopic Surgery
Brief Title: Efficacy of an Erector Spinae Plane Block in VATS/RATS
Acronym: ESPAM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UZB-VUB-19-01; 2019-003534-17 (EudraCT Number)
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Pain, Postoperative; Post-Op Complication
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Single-blinded, single-center, randomized, prospective study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- PCIA arm (No Intervention): Standard post-operative treatment with patient-controlled intravenous analgesia (Piritramide bolus = 2mg, bolus interval = 7 minutes, max 4 hour dose = 30mg)
- ESP block arm (Active Comparator): ultrasound guided Erector spinae block (Single shot of 30ml of 0.5% solution of Naropin [Ropivacaine])
  Interventions: Drug: Erector spinae plane block with ropivacaine 3.75mg/ml
- IC block arm (Active Comparator): 3 ml of 0.5% solution of Naropin [Ropivacaine] per intercostal space, up to a maximum of 30ml
  Interventions: Drug: Erector spinae plane block with ropivacaine 3.75mg/ml

INTERVENTIONS:
Drug: Erector spinae plane block with ropivacaine 3.75mg/ml — Single shot erector spinae block
  Other Names: Naropin
  Arms: ESP block arm; IC block arm

SUMMARY:
This study aims to study the analgesic and respiratory effects of the erector spinae plane block for patients undergoing video-assisted thoracic surgery (VATS) or robotic assisted thoracic surgery (RATS).

DETAILED DESCRIPTION:
A total of 120 subjects will be randomized into three groups (30 per group). Arm A: IV PCIA Arm B: IV PCIA + ultrasound guided Erector spinae block (ESPB, Single shot of 30ml of 0.5% solution of Naropin [Ropivacaine]) Arm C: IV PCIA + multilevel intra-thoracic intercostal nerve block (ICB, Single shot of 30ml of 0.5% solution of Naropin [Ropivacaine]) PCIA pumps for all study cohorts will be programmed according to our institution's standard protocol (Dipidolor [Piritramide] bolus: 2mg, interval: 7 min, max 4h dose: 30mg). The erector spinae block will be placed preoperatively, the intercostal block will be placed at the beginning of the procedure. All patients will receive standard postoperative care. The patients will be blinded for the study arm.

The primary endpoint of this study is postoperative pain and will be recorded by using the numerical rating scale (NRS) pain score. Pain scores will be measured by the investigator at rest and during coughing. Opioid consumption will be monitored and registered for.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* age between 18 to 100 years old
* ASA 1-3
* scheduled for VATS
* informed consent explained and signed

Exclusion Criteria:

* Patients < 18 years old, > 100 years old
* ASA physical status > 3
* previous cardiac surgery or ipsilateral thoracic surgery
* neuropsychiatric diseases
* allergy to analgesics or local anesthetics or other medications used in the study
* abuse of opioids or sedatives
* contraindication to receive regional anesthesia (e.g. coagulation defect)
* patients who could not understand the VAS pain-scoring system
* patient refusal to follow participation
* expected post operative mechanical ventilation
* intolerance or allergy to any prescribed medication

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-06-28 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of ESP block in decreasing postoperative pain intensity | 48 hours
  Pain levels will be assessed using the 10 points Visual analogue Scale (VAS) where zero= no pain and 10= pain as bad as it can be. The vaS is a validated tool to measure pain and discomfort. It is sensitive to pharmacological and non-pharmacological interventions, that have an impact over the experience of pain, as well as it's high correlation with pain levels

IPD SHARING:
Plan to Share IPD: No